CLINICAL TRIAL: NCT02275442
Title: Effect of Precariousness in RUral Areas During preGNANCY
Acronym: PRUGNANCY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Hospital Center of Issoire : Maternity unit (Unknown); PEPRADE label unit EA 4681 : Department of general practice - Clermont-Ferrand AND Unit of Epidemiology, economic health and prevention - C.H.U Clermont-Ferrand (Unknown); Perinatal cares Auvergne network - C.H.U Estaing, Clermont-Ferrand (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-0212
Record Dates: First submitted 2014-10-03; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Pregnancy; Rural Parturient Women; Precarious Situation; EPICES Scale; General Practice
Keywords: EPICES scale; Precarious situation; Rural parturient women; Access to care; Global Initiative for Sentinel E-health Network on Grid; General practice

INTERVENTIONS:
Other: EPICES scale

SUMMARY:
The link between precarious situations and health conditions are more described in previous study. Precarious situations are more frequent and complex especially in rural areas. There are recognized like a risk factor of complications during pregnancy and delivery. It's necessary to describe antenatal cares for rural women in precarious situations to prevent those situations, to understand their difficulties in order to reduce inequalities and health spending.

The aim of the PRUGNANCY study is to understand the difficulties of rural parturient women and the strategies developed to overcome them. Recognized earlier precarious situations and valorized General Practitioners and restore them to the follow-up or parturient women.

DETAILED DESCRIPTION:
It's a multicenter prospective observational study with a quali-quantitative method. This study involved three maternities in Auvergne region (Issoire, Thiers, Saint-Flour). Precarious women living in rural areas are included. They will be followed during a period of two months after childbirth. The main assessment criterion is the adequation rate between antenatal care for those women and the HAS recommendation's.

The amount necessary to highlight a significant difference is 190 patients (IC 95% [0.429 - 0.571] ; risk = 5 % ; Adequation rate = 50 % ; lost to follow-up rate = 10 % ; deprivation rate = 27 %).

The secondary criteria of judgment are the reasons for not realized antenatal and postnatal cares, the difficulties of realized antenatal and postnatal cares, the strategies developed to overcome them, the term and health status of the child birth (Apgar score, birth weight), the health status of the child birth and his mother during the two post-partum months (HAS recommendation's).

ELIGIBILITY:
Inclusion Criteria:

* Women old enough to procreate. Precariousness: EPICES scale > 30, 17. Live in rural areas (INSEE definition).

Exclusion Criteria:

* To be unable to answer the questionnaire: intellectual disability or no French speaker or illiterates.

EPICES scale not completed. Women who gave birth to a stillborn child. Medical interruption of pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: rural parturient women
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
rate for prenatal cares | at 9 months

SECONDARY OUTCOMES:
antenatal and postnatal cares | at day 1
strategies to overcome difficulties to realize antenatal and postanatal cares | at 2 months
  questionnaires with open-ended questions to invite further comments

CONTACTS AND LOCATIONS:
Overall Officials: Philippe VORILHON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France